CLINICAL TRIAL: NCT01373996
Title: Feasibility and Accuracy of Wireless Transmission of Invasive Blood Pressure Signal From Patient to Patient's Bedside Monitor
Brief Title: Clinical Investigation of Wireless Transmission of Invasive Blood Pressure Signal
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: Hyb, d.o.o., Slovenia (Unknown)
Responsible Party: UMC Ljubljana (Primoz Gradisek), UMC Ljubljana
Other Study IDs: HMW10
Record Dates: First submitted 2011-06-10; First posted 2011-06-15 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2011-04

CONDITIONS: Multiple Trauma; Shock; Atrial Fibrillation; Perioperative/Postoperative Complications
Keywords: Invasive blood pressure monitoring; Intensive care unit; Wireless Technology
MeSH Terms: conditions — Multiple Trauma; Shock; Atrial Fibrillation; Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Wireless: Measuring of invasive arterial blood pressure through HMW10 Wireless System.
  Interventions: Device: Wireless invasive blood pressure monitoring (Hybymed® Wireless IBPM System)
- Wired: Measuring of invasive arterial blood pressure through conventional wired technology.

INTERVENTIONS:
Device: Wireless invasive blood pressure monitoring (Hybymed® Wireless IBPM System) — The readings of invasive arterial pressure were obtained from 2 identical pressure transducers, connected to a common arterial line via a Y connector. Data was collected from one transducer via a direct cable connection and from the second transducer via wireless transmission of the signal to the patient's bedside monitor using the HMW 10 Wireless System.
  A comparison of data received by patient's bedside monitor from the two transducers was done (standard connection vs. wireless connection), as well as a comparison of data collected by the transmitter and data received by the receiver of the HMW 10 Wireless System.
  Other Names: Hybymed® Wireless IBPM System HMW10. Hyb d.o.o., Slovenia
  Groups: Wireless

SUMMARY:
The purpose of this study is to determine whether wireless transmission of invasive arterial blood pressure signal (by HMW 10 Wireless System) from patient to patient's bedside monitor is feasible, safe and as accurate as conventional cable connection.

DETAILED DESCRIPTION:
The technology for invasive arterial blood pressure measurement in emergency room, operating theater, recovery room and intensive care unit is well established and uses pressure sensor connected via cable to patient's bedside monitor. The wireless sensors result in reduction of wires attached to the patient and may enhance nursing, treatment and transportation of patients in aforementioned setting.

The HMW 10 Wireless System was developed and incorporates wireless transmission of patient's signal. The purpose of the study was to measure the quality of data transmitted through the HMW 10 Wireless System, and to demonstrate that the quality of the data meets the requirements of European Directive 93/42/EEC (Medical Device Directive - MDD) and EN/IEC 60601-1 and EN/IEC 60601-2-34.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients requiring invasive blood pressure monitoring

Exclusion Criteria:

* frequent blood sampling through arterial cannula (more than 3 times a day)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2011-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Difference between wired and wireless invasive arterial blood pressure | 24 hours of monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Primoz Gradisek, MD, Principal Investigator — UMC Ljubljana; Neva Pozar-Lukanovic, MD, MMsc, Principal Investigator — UMC Ljubljana